CLINICAL TRIAL: NCT00734110
Title: Multi-Centre Clinical Study of the P.F.C.® Sigma Total Knee System
Brief Title: Long-term Study of The Press Fit Condylar (P.F.C.) Sigma Total Knee Replacement System
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study achieved the stated objective to record pre & post operative outcomes at a minimum 5 years.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT 99/24
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis
Keywords: Arthroplasty, Replacement, Knee, P.F.C. Sigma RPF, Sigma RP
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P.F.C. Sigma Total Knee Replacement System (Experimental): Primary total knee arthroplasty using the fixed bearing P.F.C. Sigma Total Knee Replacement System.
  Interventions: Device: P.F.C. Sigma Total Knee System

INTERVENTIONS:
Device: P.F.C. Sigma Total Knee System — An orthopaedic implant for total knee replacement
  Other Names: Sigma Fixed Bearing Total Knee System

SUMMARY:
The main purpose of this study is to record information from clinical and radiographic examinations and patient assessment questionnaires before surgery and at suitable postoperative intervals to assess the functioning and symptomology of each knee following surgery.

In addition, any adverse events or complications are to be recorded, and any device failures or early revisions are to be recorded and reported directly to the Sponsor. The data are to be used in an evaluation of the performance of the P.F.C. Sigma knee implants over a minimum of 5 years.

DETAILED DESCRIPTION:
The primary outcome measures are detailed above in the brief summary. Secondary outcomes are any adverse events or complications and any device failures or early revisions to be recorded and reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given voluntary written informed consent to participate in this study.
* Patients for whom primary Total Knee Replacement is indicated due to degenerative joint disease, including rheumatoid arthritis, osteoarthritis, avascular necrosis, and post-traumatic arthritis, which is causing pain, deformity, or limitation of function uncontrolled by medical treatment.
* Patients who, in the opinion of the Investigator, are able to understand this study, co-operate with the investigational procedures and are willing to return to the hospital for all the scheduled post-operative follow-ups.
* Male or female patients who are skeletally mature and for whom an appropriate size of device is available.

Exclusion Criteria:

* Patients scheduled for Revision Total Knee Arthroplasty, or who have had previous surgery to their knee except menisectomy, arthroscopy or synovectomy.
* Patients experiencing any condition that may, in the opinion of the Investigator, interfere with the Total Knee Replacement's survival or outcome (e.g. Paget's disease, Charcot's disease, severe osteoporosis, etc.)
* Patients who have evidence of active infections which may spread to other areas of the body (e.g. osteomyelitis, pyrogenic infection of the knee joint, overt infection, etc.).
* Patients who are currently participating in any other clinical investigation of a device or pharmaceutical.
* Patients having non-contained defects in the tibia or femur necessitating bone graft.
* Patients with psychosocial disorders that would limit rehabilitation or follow-up.
* Subjects with a known history of poor compliance to medical treatment.
* Subjects who are known drug or alcohol abusers.
* Other contraindications for the use of the P.F.C. ® S Knee System as listed in the package insert.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2000-07-01 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2010-06-01 (Actual)

PRIMARY OUTCOMES:
To record information from clinical and radiographic examinations and patient assessment questionnaires before surgery and at suitable postoperative intervals | 5 years

SECONDARY OUTCOMES:
The secondary outcomes are any adverse events or complications are to be recorded, and any device failures or early revisions are to be recorded and reported. | 6 weeks, 1, 2, 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Alexandra Hospital NHS Trust, Harlow, Essex, United Kingdom